CLINICAL TRIAL: NCT00851110
Title: A Prospective Randomized Feasibility and Phase II Adjuvant Breast Cancer Study of the Netherlands Working Party for Autotransplantation in Solid Tumors.
Brief Title: Adjuvant Breast Cancer Study of the Netherlands Working Party for Autotransplantation in Solid Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METc 2004/110; CKTO 2005-15
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2009-02-25 (Estimated); Status verified 2009-02

CONDITIONS: High-Risk Breast Cancer
Keywords: high dose; breast cancer; adjuvant
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy

INTERVENTIONS:
Procedure: stem cell reinfusion — hematopoietic stem cell reinfusion
Drug: Chemotherapy — High-dose chemotherapy consisting of cyclophosphamide, thiotepa and carboplatin

SUMMARY:
Objectives of the study:

This randomized multicenter phase II study compares the tolerability, toxicity and quality of life between two high-dose chemotherapy regimens based on cyclophosphamide, thiotepa and carboplatin.

Regimen A: full dose CTC. Regimen B: two courses of CTC (tCTC) with 33% dose reduction.

Primary endpoints are:

* Maximum degree of non-hematological toxicity.

Secondary endpoint:

* Total number of hospital days.
* Quality of life evaluations during and following high-dose chemotherapy (up to 1 year).
* Effect of therapeutic dose monitoring of CTC or tCTC.

Trial design:

This investigation is a multicenter prospective randomized phase II study. Patients eligible for the study will be identified after mastectomy or wide tumor excision with axillary clearance. Following randomization, all patients will receive four courses of cyclophosphamide, epirubicin and fluorouracil (FEC). Patients with early progressive disease at any time will be taken off study. The first chemotherapy course must be given as soon as possible after the surgical procedure, preferably within 3 weeks, but not later than 6 weeks since primary surgery. After the third or fourth FEC course G-CSF is administered and peripheral stem cells will be harvested. All radiation therapy (including radiation therapy administered as part of a breast conserving strategy) must be postponed until all chemotherapy has been concluded.

Questionnaires, comprising the Rotterdam Symptom Checklist (RSCL) and the Short-Form General Health Survey (SF-36) will be sent by mail before randomization, after chemotherapy, 3 months thereafter, further on every l/2 yr till at least 1 year follow-up as performed earlier. [6, 28, 29].

All patients will be randomized before the initiation of chemotherapy.

* The 'standard' treatment arm will include 4 courses of FEC followed by high-dose chemotherapy with a single course of full dose CTC followed by peripheral stem cell reinfusion. Subsequently, conventional external beam radiotherapy to the breast or chest wall and to the regional lymph node areas including the axilla and the parasternal area will be administered following guidelines of the individual center. Patients with hormone receptor positive disease will go on to receive 5 years of tamoxifen. Patients with receptor positive disease who have not entered menopause will be advised to undergo ovarian ablation as well.
* The 'experimental' treatment arm will be identical to the 'standard' one, except that the single course of CTC will be replaced by 2 courses of tCTC each followed by peripheral stem cell reinfusion.

DETAILED DESCRIPTION:
High-dose chemotherapy with the alkylating agent combination CTC appears to add significantly to the efficacy of conventional dose chemotherapy in patients with high-risk breast cancer, provided that the HER-2/neu gene is not amplified in the tumor. As a high-dose chemotherapy regimen, CTC is associated with significant toxicity [31,32]. Although high-dose alkylating therapy seems to be effective, there is virtually nothing known about the dose-response curve for this combination (for a detailed discussion see the classical paper by E. Frei III [32]. If one assumes that the efficacy increase levels off with increasing dose, the efficacy of tCTC might be almost as great as that of CTC, but with considerably less toxicity. In addition, two closely spaced courses of tCTC might further increase the efficacy of the regimen. There are some suggestions that a double transplant may be more effective than a single one, in multiple myeloma and in Ewing sarcoma. A similar suggestion has also been made for breast cancer (study of Nitz et al ref 4, table 1).

ELIGIBILITY:
Inclusion criteria:

1. Modified radical mastectomy (or breast conserving surgery) and axillary clearance, histologically confirmed stage IIA, IIB or IIIA adenocarcinoma (excluding supraclavicular lymph nodes) of the breast, with 4 or more involved axillary lymph nodes. Presence of tumor cells near or in the resection margins at microscopic examination is acceptable
2. The primary tumor must be immunohistochemically negative for HER-2/neu expression. An immunohistochemistry score of 1+ is also acceptable. A score of 3+ is not acceptable. A score of 2+ is only acceptable if a FISH analysis (or equivalent) has clearly shown that there is no HER-2/neu gene-amplification
3. No prior chemotherapy or radiotherapy
4. No evidence of distant metastases
5. Age < 50 years
6. Performance status (ECOG-ZUBROD) 0 or 1;
7. Normal bone marrow function, WBC > 4.0 x 109/l, platelets > 100 x 109/l;
8. Adequate renal function (creatinine clearance > 60 ml/min.);
9. Adequate hepatic function (serum bilirubin < 25 umol/l);
10. Study treatment must begin within 6 weeks of surgery;
11. No other malignancy except adequately treated in situ carcinoma of the cervix or basal cell carcinoma of the skin;
12. No significant prior or concomitant disorder that might interfere with adherence to the intensive treatment regimen, including but not limited to a history of angina, myocardial infarction or heart failure, severe lung function impairment, peptic ulcer disease, etc.;
13. Availability for follow-up.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-10

PRIMARY OUTCOMES:
Maximum degree of non-hematological toxicity.

SECONDARY OUTCOMES:
Total number of hospital days
Quality of life evaluations during and following high-dose chemotherapy (up to 1 year)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth G.E. de Vries, MD, PhD, Study Director — University Medical Center Groningen; Sjoerd Rodenhuis, MD, PhD, Study Director — The Netherlands Cancer Institute
Locations (10):
- Netherlands (10):
  - Free University Hospital, Amsterdam
  - The Netherlands Cancer Institute, Amsterdam
  - Academic Medical Center, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - University Medical Centre Groningen, Groningen
  - Leiden University Medical Centre, Leiden
  - University Hospital Maastricht, Maastricht
  - University Medical Centre Nijmegen St. Radboud, Nijmegen
  - Erasmus MC, Daniel den Hoed Cancer Center, Rotterdam
  - University Medical Centre Utrecht, Utrecht

REFERENCES:
- [Background] Weiss RB, Rifkin RM, Stewart FM, Theriault RL, Williams LA, Herman AA, Beveridge RA. High-dose chemotherapy for high-risk primary breast cancer: an on-site review of the Bezwoda study. Lancet. 2000 Mar 18;355(9208):999-1003. doi: 10.1016/S0140-6736(00)90024-2. PMID 10768448
- [Background] Bergh J, Wiklund T, Erikstein B, Lidbrink E, Lindman H, Malmstrom P, Kellokumpu-Lehtinen P, Bengtsson NO, Soderlund G, Anker G, Wist E, Ottosson S, Salminen E, Ljungman P, Holte H, Nilsson J, Blomqvist C, Wilking N. Tailored fluorouracil, epirubicin, and cyclophosphamide compared with marrow-supported high-dose chemotherapy as adjuvant treatment for high-risk breast cancer: a randomised trial. Scandinavian Breast Group 9401 study. Lancet. 2000 Oct 21;356(9239):1384-91. doi: 10.1016/s0140-6736(00)02841-5. PMID 11052580
- [Background] Tallman MS, Gray R, Robert NJ, LeMaistre CF, Osborne CK, Vaughan WP, Gradishar WJ, Pisansky TM, Fetting J, Paietta E, Lazarus HM. Conventional adjuvant chemotherapy with or without high-dose chemotherapy and autologous stem-cell transplantation in high-risk breast cancer. N Engl J Med. 2003 Jul 3;349(1):17-26. doi: 10.1056/NEJMoa030684. PMID 12840088
- [Background] Nitz UA, Frick M, Mohrmann S. Lindemann H, Jackisch C, Werner C, Souchon R, Metzner B, Rufert U, Bender HG. Tandem high dose chemotherapy versus dose-dense conventional chemotherapy for patients with high risk breast cancer: Interim results from a multicenter phase III trial. Proc Am Soc Clin Oncol 22: 2003 (abstract 3344).
- [Background] Servent V, Bonneterre J, Roche H, Kerbrat P, Bremond A, Fumoleau P, Namer M, Goudier MJ, Fargeot P, Chapelle-Marcillac I. 10-year follow-up update of French adjuvant study gropu 05 trial: FEC 100 regimen remains superior to FEC 50 in adjuvant chemotherapy of poor prognosis, node-positive, early breast cancer patients. Breast 12 Suppl 1: S35, 2003.
- [Background] Rodenhuis S, Bontenbal M, Beex LV, Wagstaff J, Richel DJ, Nooij MA, Voest EE, Hupperets P, van Tinteren H, Peterse HL, TenVergert EM, de Vries EG; Netherlands Working Party on Autologous Transplantation in Solid Tumors. High-dose chemotherapy with hematopoietic stem-cell rescue for high-risk breast cancer. N Engl J Med. 2003 Jul 3;349(1):7-16. doi: 10.1056/NEJMoa022794. PMID 12840087
- [Background] Peters WP, Rosner G, Vredenburgh J, Shpall EJ, Crump M, Marks L, Cirrincione C, Hurd D, Norton L, Ann B. Updated results of a prospective, randomized comparison of two doses of combination alkyating agents (AA) as consolidation after CAF in high-risk primary breast cancer involving ten or more axillary lymph nodes (LN): CALGB 9082/SWOG 9114/NCIC Ma-13. Proc ASCO 20:81, 2001
- [Background] Gianni A, Bonadonna G. Five-Year Results of the randomized clinical trial comparing standard versus high-dose myeloablative chemotherapy in the adjuvant treatment of breast cancer with > 3 positive nodes (LN+). Proc ASCO 20: 80, 2001
- [Background] Rodenhuis S, Westermann A, Holtkamp MJ, Nooijen WJ, Baars JW, van der Wall E, Slaper-Cortenbach IC, Schornagel JH. Feasibility of multiple courses of high-dose cyclophosphamide, thiotepa, and carboplatin for breast cancer or germ cell cancer. J Clin Oncol. 1996 May;14(5):1473-83. doi: 10.1200/JCO.1996.14.5.1473. PMID 8622061
- [Background] Rodenhuis S, de Wit R, de Mulder PH, Keizer HJ, Sleijfer DT, Lalisang RI, Bakker PJ, Mandjes I, Kooi M, de Vries EG. A multi-center prospective phase II study of high-dose chemotherapy in germ-cell cancer patients relapsing from complete remission. Ann Oncol. 1999 Dec;10(12):1467-73. doi: 10.1023/a:1008328012040. PMID 10643538
- [Background] Rodenhuis S, Demol J, Westermann A, Holtkamp MJ, Nooijen WJ, Slaper-Cortenbach ICM, Schornagel JH, Baars JW: The feasibility of three courses of 'tiny CTC' (tCTC) in patients with advanced breast cancer. in: KA Dicke and A Keating (Eds.) Autologous Marrow and Blood Transplantation. Proceedings of the Eighth International Symposium Arlington, Texas. Carden Jennings Publishing Company, Charlottesville, Virginia 1997. p 277-285
- [Background] Schrama JG, Baars JW, Holtkamp MJ, Schornagel JH, Beijnen JH, Rodenhuis S. Phase II study of a multi-course high-dose chemotherapy regimen incorporating cyclophosphamide, thiotepa, and carboplatin in stage IV breast cancer. Bone Marrow Transplant. 2001 Jul;28(2):173-80. doi: 10.1038/sj.bmt.1703105. PMID 11509935
- [Background] Westermann AM, Holtkamp MM, Linthorst GA, van Leeuwen L, Willemse EJ, van Dijk WC, Nooijen WJ, Baars JW, Schornagel JH, Rodenhuis S. At home management of aplastic phase following high-dose chemotherapy with stem-cell rescue for hematological and non-hematological malignancies. Ann Oncol. 1999 May;10(5):511-7. doi: 10.1023/a:1026427724108. PMID 10415999
- [Background] van Warmerdam LJ, Rodenhuis S, van Tellingen O, Maes RA, Beijnen JH. Validation of a limited sampling model for carboplatin in a high-dose chemotherapy combination. Cancer Chemother Pharmacol. 1994;35(2):179-81. doi: 10.1007/BF00686644. PMID 7987998
- [Background] van Warmerdam LJ, Rodenhuis S, van der Wall E, Maes RA, Beijnen JH. Pharmacokinetics and pharmacodynamics of carboplatin administered in a high-dose combination regimen with thiotepa, cyclophosphamide and peripheral stem cell support. Br J Cancer. 1996 Apr;73(8):979-84. doi: 10.1038/bjc.1996.191. PMID 8611435
- [Background] van Maanen RJ, van Ooijen RD, Zwikker JW, Huitema AD, Rodenhuis S, Beijnen JH. Determination of N,N',N"-triethylenethiophosphoramide and its active metabolite N,N',N"-triethylenephosphoramide in plasma and urine using capillary gas chromatography. J Chromatogr B Biomed Sci Appl. 1998 Nov 20;719(1-2):103-12. doi: 10.1016/s0378-4347(98)00381-8. PMID 9869370
- [Background] van Maanen MJ, Tijhof IM, Damen JM, Versluis C, van den Bosch JJ, Heck AJ, Rodenhuis S, Beijnen JH. A search for new metabolites of N,N',N''-triethylenethiophosphoramide. Cancer Res. 1999 Sep 15;59(18):4720-4. PMID 10493531
- [Background] van Maanen MJ, Huitema AD, Rodenhuis S, Beijnen JH. Urinary excretion of thioTEPA and its metabolites in patients treated with high-dose cyclophosphamide, thioTEPA and carboplatin. Anticancer Drugs. 2001 Jul;12(6):519-24. doi: 10.1097/00001813-200107000-00005. PMID 11459998
- [Background] Huitema AD, Tibben MM, Kerbusch T, Kettenes-van den Bosch JJ, Rodenhuis S, Beijnen JH. Simple and selective determination of the cyclophosphamide metabolite phosphoramide mustard in human plasma using high-performance liquid chromatography. J Chromatogr B Biomed Sci Appl. 2000 Aug 18;745(2):345-55. doi: 10.1016/s0378-4347(00)00295-4. PMID 11043753
- [Background] Huitema ADR, Tibben MM, Kerbusch T, Kettenes-van den Bosch JJ, Rodenhuis S, Beijnen JH: High performance liquid chromatographic determination of the stabilized cyclophosphamide metabolite 4-hydroxycyclophosphamide in plasma and red blood cells. J Liq Chrom Rel Technol 2000, 23: 1725-1744
- [Background] Huitema AD, Reinders C, Tibben MM, Rodenhuis S, Beijnen JH. Sensitive gas chromatographic determination of the cyclophosphamide metabolite 2-dechloroethylcyclophosphamide in human plasma. J Chromatogr B Biomed Sci Appl. 2001 Jun 15;757(2):349-57. doi: 10.1016/s0378-4347(01)00178-5. PMID 11417881
- [Background] Huitema ADR, Mathôt RAA, Tibben MM, Reinders C, Rodenhuis S, Beijnen JH: Pharmacokinetics of cyclophosphamide and its metabolite 2-dechloroethylcyclophosphamide in a high-dose combination with thioTEPA and carboplatin. Submitted
- [Background] Huitema AD, Kerbusch T, Tibben MM, Rodenhuis S, Beijnen JH. Reduction of cyclophosphamide bioactivation by thioTEPA: critical sequence-dependency in high-dose chemotherapy regimens. Cancer Chemother Pharmacol. 2000;46(2):119-27. doi: 10.1007/s002800000132. PMID 10972481
- [Background] Huitema AD, Mathot RA, Tibben MM, Rodenhuis S, Beijnen JH. A mechanism-based pharmacokinetic model for the cytochrome P450 drug-drug interaction between cyclophosphamide and thioTEPA and the autoinduction of cyclophosphamide. J Pharmacokinet Pharmacodyn. 2001 Jun;28(3):211-30. doi: 10.1023/a:1011543508731. PMID 11468938
- [Background] Schrama JG, Holtkamp MJ, Baars JW, Schornagel JH, Rodenhuis S. Toxicity of the high-dose chemotherapy CTC regimen (cyclophosphamide, thiotepa, carboplatin): the Netherlands Cancer Institute experience. Br J Cancer. 2003 Jun 16;88(12):1831-8. doi: 10.1038/sj.bjc.6601001. PMID 12799623
- [Background] Frei E 3rd, Antman K, Teicher B, Eder P, Schnipper L. Bone marrow autotransplantation for solid tumors--prospects. J Clin Oncol. 1989 Apr;7(4):515-26. doi: 10.1200/JCO.1989.7.4.515. PMID 2647915
- [Background] ten Vergert EM, S Rodenhuis, M Bontenbal, DJ Richel, JH Schornagel, NH Mulder, J Wagstaff, CJ Rodenburg, GH Blijham, de Wit R, MA Nooy, LV Beex, PS Hupperets, de Vries EG. Quality of life in a randomized adjuvant breast carcinoma study with standard vs high dose chemotherapy Proc Am Soc Clin Oncol. Abstract No: 77 1996
- [Background] Buijs C, Nieboer P, Rodenhuis S, Bontenbal M, Van der Wall E, Nooij MA, Voest EE, Ten Vergert EM, Mulder NH, Van der Graaf WTA. Fatigue after adjuvant chemotherapy for breast cancer.Proc Am Soc Clin Oncol 22: Abstract No: 127, 2003
- [Background] Hematopoietische stamcellen.Gezondheidsraad. Den Haag: Gezondheidsraad, 2003; publicatie nr 2003/17. ISBN: 90-554-497-6
- [Background] Miller JS, Arthur DC, Litz CE, Neglia JP, Miller WJ, Weisdorf DJ. Myelodysplastic syndrome after autologous bone marrow transplantation: an additional late complication of curative cancer therapy. Blood. 1994 Jun 15;83(12):3780-6. PMID 8204897
- [Background] Neglia J, Shapiro R, Haake R, Ramsay N, McGlave P, Kersey J. Bone marrow transplantation-II. Allogeneic transplantation-clinical studies. Second neoplasms (SNs) following bone marrow transplantation (BMT) [Abstract 667]. Blood 80, 1992
- [Background] Manual for Clinical Research a Breast Cancer by the EORTC Breast Cancer Cooperative Group, Leuven, 1991
- [Background] Quality assurance in conservative treatment of early breast cancer, a consensus meeting. December 13-14, 1990, Tubingen, Germany. Radiother Oncol. 1991 Dec;22(4):219-338. No abstract available. PMID 1792309
- [Background] Goss PE, Ingle JN, Martino S, Robert NJ, Muss HB, Piccart MJ, Castiglione M, Tu D, Shepherd LE, Pritchard KI, Livingston RB, Davidson NE, Norton L, Perez EA, Abrams JS, Therasse P, Palmer MJ, Pater JL. A randomized trial of letrozole in postmenopausal women after five years of tamoxifen therapy for early-stage breast cancer. N Engl J Med. 2003 Nov 6;349(19):1793-802. doi: 10.1056/NEJMoa032312. Epub 2003 Oct 9. PMID 14551341